CLINICAL TRIAL: NCT06089551
Title: Early Versus Postponed Supplementary Parenteral Nutrition After Major Emergency Abdominal Surgery: A Randomized, Controlled Multicenter Trial
Brief Title: Early vs Postponed Parenteral Nutrition After Emergency Abdominal Surgery
Acronym: EATERS
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Copenhagen University Hospital at Herlev (Other)
Collaborators: Copenhagen University Hospital, Hvidovre (Other); Nordsjaellands Hospital (Other); Slagelse Sygehus (Other); Aarhus University Hospital (Other); Gødstrup Hospital (Other); Aalborg University Hospital (Other); Bispebjerg Hospital (Other); Zealand University Hospital (Other); Holbaek Sygehus (Other)
Responsible Party: Principal Investigator, Jannick Brander Hansen, Principal Investigator, Copenhagen University Hospital at Herlev
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: The EATERS Trial
Record Dates: First submitted 2023-09-26; First posted 2023-10-18 (Actual); Last update posted 2025-02-12 (Actual); Status verified 2024-02

CONDITIONS: Laparotomy; Bowel Obstruction; Ischemia, Mesenteric
Keywords: Major emergency laparotomy; Supplementary parenteral nutrition
MeSH Terms: conditions — Intestinal Obstruction; Mesenteric Ischemia

STUDY DESIGN:
Intervention Model Description: Randomized study with two study groups
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Early supplementary (Experimental): Start of study drug on postoperative day 2
  Interventions: Drug: SmofKabiven
- Late supplementary (Active Comparator): Start of study drug on postoperative day 5
  Interventions: Drug: SmofKabiven

INTERVENTIONS:
Drug: SmofKabiven — Participants will receive supplementary parenteral nutrition based on their calorie intake. The dosage will be adjusted on a daily basis depending on intake.
  Other Names: SmofKabiven Perifer

SUMMARY:
The aim of this study is to investigate the effect of early, supplementary parenteral nutrition following emergency laparotomy.

Currently, parenteral nutrition is used in postoperative patients if or when oral or enteral nutrition is not feasible. However, little data exists on the optimal timing of parenteral nutrition.

Oral and enteral nutrition is encouraged. Participants will randomized on the second postoperative day if their calorie intake (oral + enteral) is below 50% of the calculated requirement. Patients will be randomized to early (postoperative day 2) or postponed (postoperative day 5) start of parenteral nutrition.

The combined oral + enteral + parenteral calorie target is 70-80% of the calculated requirement. Participants in the postponed group will be re-assessed on postoperative day 5, and if their calorie intake is less than 50% parenteral nutrition will be administered.

The intervention will continue until oral + enteral intake is at least 70% of the calculated requirement or the participant is at his/her habitual intake.

DETAILED DESCRIPTION:
Screening for potential participants will be done using the patient records which includes primary procedure, age, NRS-2002 score, and total calorie intake within the last 24 hours. Only information needed to determine eligibility in this study will be noted ahead of informed consent.

Enteral or oral feeding is encouraged as soon as possible postoperatively for all patients unless they have contraindications for oral intake. If they have contraindications for oral intake they are excluded from participation (Appendix 2). The caloric target is set to 25 kcal/kg/day. For patients with a body mass index > 30 kg/m2 the target will be calculated using their weight at body mass index 25 kg/m2. Oral protein supplements are encouraged in all patients. Nutritional calculations and monitoring can be performed locally according to the participating centers' standard clinical practice by dieticians, nurses, or clinical doctors.

Patients that cannot achieve more than 50% of their calorie intake on POD2 and do not fulfill any of the exclusion criteria are randomized to early parenteral (E-SPN) (POD2) or postponed parenteral (L-SPN) (POD5). The L-SPN group will continue standard oral or enteral intake until POD5 where the parenteral nutritional intervention begins if they have not yet met at least 50% of recommended daily oral or enteral recommended intake on their own.

After randomization, the patients should receive 70-80% of recommended daily energy and protein intake. Calculations will be made daily by a combination of oral, enteral, and parenteral administered nutrition. In case of incomplete calorie intake registration, the most recent dose will be administered.

If patients are in need of supplemental parenteral nutrition for more than seven days, a centrally administered route should be used. The standard trial supplemental nutritional product will be SmofKabiven® Perifer unless there is a clinical rationale for using SmofKabiven. These include treatment duration > 7 days, risk of overhydration, calorie requirement exceeding the limit for SmofKabiven Perifer (1300 kcal). Both products will be used in accordance with the summary of product characteristics. Use of either product is not expected to impact data analysis as supplementary calorie amount is unrelated to the product.

Both investigational medicinal products (IMP) will be supplied by the local hospital pharmacy. All IMPs are stored in a dedicated medicine storage room located on each hospital ward. Handling IMPs will be in accordance with the regional guideline on the use of parenteral nutrition (Parenteral ernæring for voksne - procedure og forholdsregler, section 3 - vip.regionh.dk). The dosage is evaluated daily and is documented in the patient chart in Sundhedsplatformen (Epic Systems Corporation, Verona, Wisconsin) as is the time of infusion start.

Batch number and expiration date will be registered on a worksheet along with the end-infused dose. Worksheets will be stored in the Trial Master File.

Destruction of the IMP will be in accordance with local standards.

Patients will be monitored regarding complications, nutritional intake (calories, protein, lipids), and safety parameters (risk of overfeeding and refeeding) as standard.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18
* Emergency primary midline laparotomy or laparoscopy
* NRS-2002 (nutritional risk screening) score < 7
* No contraindications for oral or enteral nutrition after surgery
* Unable to tolerate or take in at least 50% of calculated calorie requirement on postoperative day 2
* Capable of providing informed consent at the time of inclusion

Exclusion Criteria:

* Laparotomy without closure of the abdominal aponeurosis
* Laparoscopic appendectomy or cholecystectomy as the procedure
* Limiting mental or psychiatric disorders rendering participation unethical or unrealistic
* Patients with a very limited expected remaining time of living (< 3 months)
* NRS-2002 = 7
* Pregnant or breastfeeding women
* Refusal to participate

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 342 (Estimated)
Dates: Start 2023-10-18 (Actual); Primary Completion 2025-10-25 (Estimated); Study Completion 2026-01-01 (Estimated)

PRIMARY OUTCOMES:
Infectious complications during admission | 1 week after hospital discharge
  Rate of infectious complications during admission. The following infections will be registered: Urinary tract infections, pneumonia, bloodstream infections, surgical site infections, abdominal infections, and skin and soft tissue infections,

SECONDARY OUTCOMES:
Non-infectious complication rate during admission | 1 week after hospital discharge
  Stratified by type and severity (Clavien-Dindo classification)
Days with need for antibiotics | 1 week after hospital discharge
  Days the participant received antibiotic treatment
Length of stay | Up to 30 days
  Time from admission to discharge
Mortality rate (day 30 and 90) | Assessed 90 days after surgery
  Mortality at day 30 and 90
Emergency readmission rate (day 30 and 90) | Assessed 90 days after surgery
  Has the participant been re-admitted within 30 or 90 days after surgery
Post-discharge nutritional status | Assessed at day 30 and 90 after surgery
  SNAQ (Simplified Nutritional Appetite Questionnaire) screening tool and weight at day 30 and 90. A score between 5 and 20 is possible with a higher score being better.
Post-discharge weight status | Assessed at day 30 and 90 after surgery
  Weight at day 30 and 90
Routes of energy delivery | Up to two weeks
  Oral intake, enteral intake, parenteral intake or a combination of the three
Energy intake during admission | Up to two weeks
  Measured in calories
Protein intake during admission | Up to two weeks
  Measured in grams of protein

CONTACTS AND LOCATIONS:
Overall Officials: Jannick B Hansen, M.D., Principal Investigator — Copenhagen University Hospital at Herlev
Locations (1):
- Herlev Hospital, Herlev, Denmark

IPD SHARING:
Plan to Share IPD: No
IPD will not be share as per Danish Law and The Data Data Protection Agency